CLINICAL TRIAL: NCT07118098
Title: INNODIA Family & Friends Early-Stage T1D Detection Protocol
Acronym: INNODIA DETECT
Status: Recruiting | Type: Observational
Sponsor: INNODIA iVZW (Other)
Responsible Party: Sponsor
Other Study IDs: INNODIA DETECT 01
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-08

CONDITIONS: Type 1 Diabetes (T1D); Pre Diabetes
Keywords: Type 1 diabetes; Autoantibodies; Screening; Pre-T1D; Stage 1; Stage 2
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Glucose Intolerance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Family and friends of people with Type 1 diabetes: Individuals with a first-degree relative with T1D have a 15-fold higher relative lifetime risk of T1D compared to the general population. Prevalence of T1D amongst individuals with a first-degree relative is 5% by age 20 compared to ~0.3% amongst the general population [10-12]. Siblings of People with T1D have, on average, a 6-7% lifetime risk of T1D, and offspring of mothers and fathers with T1D have a 1.3-4% and 6-9% lifetime risk, respectively, compared with 0.4% in the general population. The aim of the INNODIA DETECT protocol is to develop a system for identifying people at-risk and with presymptomatic T1D through targeted testing of relatives and friends of people living with symptomatic T1D. Individual will have a blood sample taken and tested for the presence of T1D autoantibodies

SUMMARY:
The purpose of INNODIA DETECT is to identify people who are at increased risk of developing T1D. Investigators are doing this by testing for markers in the blood (autoantibodies) that tell them an individuals risk of getting T1D in the future.

What is Type 1 Diabetes (T1D)? T1D is a serious disease where the blood glucose (sugar) level is too high because the body cannot make a hormone called insulin.

This happens when the body's immune system attacks the cells in the pancreas that make insulin (called beta cells), meaning that insulin production stops.

This is harmful to the body as insulin does an essential job. It allows the glucose in the blood to enter cells and fuel the body, resulting in a lowering of the blood glucose level.

What are Autoantibodies? T1D autoantibodies are markers found in the blood that indicate that the destruction of insulin producing cells has begun. The risk of developing T1D increases with the number of autoantibodies detected.

People who have 1 autoantibody detected in their blood are at increased risk of developing T1D. The presence of 2 or more autoantibodies indicates that T1D is present but the individual does not show any signs or symptoms yet.

However, these autoantibodies can be present for many years before someone develops symptoms of T1D. They often appear in the first few years of life.

The investigators are asking children and adults across Europe, aged between 1 and 45 years, who have either a family member (parent, child, full or half sibling) or close friend diagnosed with T1D before 45 years of age to provided a small blood sample so they can look at these T1D autoantibodies.

If a participant's autoantibody results are negative, this means they do not have autoantibodies and are at low risk of developing T1D. No further tests will be required, and they will exit the program.

If results indicate a participant has 1 or more positive T1D autoantibodies, a member of the clinical team will contact and invite them to the hospital for a venous blood sample to confirm the result. This confirmation test will be done as part of routine clinical care by the participants clinical team. INNODIA DETECT will end here and, if confirmed positive, the participant will be invited to attend further follow-up by entering in a separate protocol (named INNODIA MONITOR).

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent to participate
2. Be aged between 1 and 45 years
3. Have a family relative with T1D or close friend diagnosed with symptomatic T1D at age <45 years

Exclusion Criteria:

1. Previous diagnosis of stage 3 T1D or other forms of diabetes
2. Unable/unwilling to consent to participation

Ages: 1 Year to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Family and friends of people living with type 1 Diabetes. People with autoimmune disorders are of particular interest
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Presence of one or more T1D IAb | End of 2027
  Blood sample will be tested for anti-GAD, anti-IA-2, anti-insulin, and anti-ZnT8,

CONTACTS AND LOCATIONS:
Locations (5):
- Katholieke Universiteit Leuven, Leuven, Belgium
- Institut National de la Santé et de la Recherche Médicale, Paris, France
- San Raffaele Hospital, Milan, Italy
- Medical University of Silesia, Katowice, Poland
- University Medical Center Ljubljana, Ljubljana, Slovenia

REFERENCES:
- See also: INNODIA is made of professionals with various disciplinary skills and a community of expert people and families living with type 1 diabetes working together with one common focus: contribute to creating a world free of type 1 diabetes — https://www.innodia.org/innodias-clinical-trials/innodia-early-t1d-detection